CLINICAL TRIAL: NCT05624177
Title: Colonisation Efficacy of a Probiotic Chewing Gum.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BLIS Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BLTCT2022/7
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases | interventions — Mastication

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups consuming chewing gum containing Streptococcus salivarius M18.
  Group A: Probiotic Streptococcus salivarius M18 chewing gum (dose: 1 billion colony forming units per gum tablet) and chew for 5 minutes duration.
  Group B: Probiotic Streptococcus salivarius M18 chewing gum (dose: 1 billion colony forming units per gum tablet) and chew for 10-20 minutes
Who Masked: Investigator
Masking Description: A Staff member, not part of the study group will be assigned to distribute blinded samples. The investigator will not be are of the dose groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Streptococcus salivarius M18 probiotic 1 billion colony forming units chewing gum: Chew 5 minutes (Active Comparator): Streptococcus salivarius M18 chewing gum 1 billion cfu chewing the gum for 5 minutes duration.
  Interventions: Dietary Supplement: Streptococcus salivarius M18 probiotic 1 billion colony forming units chewing gum (chew 5 minutes)
- Streptococcus salivarius M18 probiotic 1 billion colony forming units chewing gum: Chew 10 minutes (Active Comparator): Streptococcus salivarius M18 chewing gum 1 billion cfu chewing the gum for 10 minutes duration.
  Interventions: Dietary Supplement: Streptococcus salivarius M18 probiotic 1 billion colony forming units chewing gum (chew 10 minutes)

INTERVENTIONS:
Dietary Supplement: Streptococcus salivarius M18 probiotic 1 billion colony forming units chewing gum (chew 5 minutes) — Probiotic Streptococcus salivarius M18 products are commercially available in traditional formats such as a chewable tablet (lozenge) for local delivery to the oral cavity to provide health benefits. In this study, a chewing gum formulation will be evaluated for its potential of delivering probiotic Streptococcus salivarius M18 to the oral cavity.
  Arms: Streptococcus salivarius M18 probiotic 1 billion colony forming units chewing gum: Chew 5 minutes
Dietary Supplement: Streptococcus salivarius M18 probiotic 1 billion colony forming units chewing gum (chew 10 minutes) — Probiotic Streptococcus salivarius M18 products are commercially available in traditional formats such as a chewable tablet (lozenge) for local delivery to the oral cavity to provide health benefits. In this study, a chewing gum formulation will be evaluated for its potential of delivering probiotic Streptococcus salivarius M18 to the oral cavity.
  Arms: Streptococcus salivarius M18 probiotic 1 billion colony forming units chewing gum: Chew 10 minutes

SUMMARY:
To evaluate the colonization efficacy (the ability of a probiotic bacteria to remain in the mouth) delivered in a chewing gum format. The chewing gum contains Streptococcus salivarius probiotic and the study is to be done in health adults.

DETAILED DESCRIPTION:
This is a single blind, randomized controlled study to evaluate the colonization effectiveness of a chewing gum containing a commercially available probiotic bacterium. Participants will be randomly assigned to one of the two groups consuming chewing gum containing Streptococcus salivarius M18 over a 7-day period. Saliva samples will be collected at pre determined points (pre and post intervention). Colonization efficacy will be determined by enumerating the probiotic from the saliva samples using standard microbiological techniques.

ELIGIBILITY:
Inclusion Criteria:

* In general, good health
* Practice good oral hygiene

Exclusion Criteria:

* Have a history of autoimmune disease or are immune compromised.
* Are on concurrent antibiotic therapy, or regular antibiotic use within last one week
* People with allergies or sensitivities to dairy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in Microbial colonization from baseline (Day 0) to 1 hour. | 1 hour post intervention.
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 chewing gum after two different times of chewing (5 vs 10 minutes). The statistical analysis will be carried out to compare the participants saliva data from baseline to post 1 hour across two different times of chewing exposure with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software.
Change in Microbial colonization from baseline (Day 0) to 8 hours. | 8 hours post intervention.
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 chewing gum after two different times of chewing (5 vs 10 minutes). The statistical analysis will be carried out to compare the participants saliva data from baseline to post 8 hours across two different times of chewing exposure with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software.
Change in Microbial colonization from baseline (Day 0) to 8 hours post last dose. | 8 hours past last dose following 7 days of twice daily administration of probiotic.
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 chewing gum after two different times of chewing (5 vs 10 minutes). The statistical analysis will be carried out to compare the participants saliva data from baseline to post 8 hours following twice daily administration of probiotic, across two different times of chewing exposure with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software.
Change in Microbial colonization from baseline (Day 0) to 48 hours post last dose. | 48 hours past last dose following 7 days of twice daily administration of probiotic.
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 chewing gum after two different times of chewing (5 vs 10 minutes). The statistical analysis will be carried out to compare the participants saliva data from baseline to post 48 hours following twice daily administration of probiotic, across two different times of chewing exposure with a level of significance of p<0.05. Overall colonization based on percentage of population colonized for different interventions will also be analyzed using appropriate statistical analysis software.

CONTACTS AND LOCATIONS:
Locations (1):
- Blis Technologies Ltd, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hyink O, Wescombe PA, Upton M, Ragland N, Burton JP, Tagg JR. Salivaricin A2 and the novel lantibiotic salivaricin B are encoded at adjacent loci on a 190-kilobase transmissible megaplasmid in the oral probiotic strain Streptococcus salivarius K12. Appl Environ Microbiol. 2007 Feb;73(4):1107-13. doi: 10.1128/AEM.02265-06. Epub 2006 Dec 28. PMID 17194838
- [Background] Burton JP, Chilcott CN, Wescombe PA, Tagg JR. Extended Safety Data for the Oral Cavity Probiotic Streptococcus salivarius K12. Probiotics Antimicrob Proteins. 2010 Oct;2(3):135-44. doi: 10.1007/s12602-010-9045-4. PMID 26781236
- [Background] Bardellini E, Amadori F, Gobbi E, Ferri A, Conti G, Majorana A. Does Streptococcus Salivarius Strain M18 Assumption Make Black Stains Disappear in Children? Oral Health Prev Dent. 2020 Apr 3;18(2):161-164. doi: 10.3290/j.ohpd.a43359. PMID 32099975
- [Background] Burton JP, Drummond BK, Chilcott CN, Tagg JR, Thomson WM, Hale JDF, Wescombe PA. Influence of the probiotic Streptococcus salivarius strain M18 on indices of dental health in children: a randomized double-blind, placebo-controlled trial. J Med Microbiol. 2013 Jun;62(Pt 6):875-884. doi: 10.1099/jmm.0.056663-0. Epub 2013 Feb 28. PMID 23449874
- [Background] Gregori G, Righi O, Risso P, Boiardi G, Demuru G, Ferzetti A, Galli A, Ghisoni M, Lenzini S, Marenghi C, Mura C, Sacchetti R, Suzzani L. Reduction of group A beta-hemolytic streptococcus pharyngo-tonsillar infections associated with use of the oral probiotic Streptococcus salivarius K12: a retrospective observational study. Ther Clin Risk Manag. 2016 Jan 19;12:87-92. doi: 10.2147/TCRM.S96134. eCollection 2016. PMID 26855579
- [Background] Di Pierro F, Adami T, Rapacioli G, Giardini N, Streitberger C. Clinical evaluation of the oral probiotic Streptococcus salivarius K12 in the prevention of recurrent pharyngitis and/or tonsillitis caused by Streptococcus pyogenes in adults. Expert Opin Biol Ther. 2013 Mar;13(3):339-43. doi: 10.1517/14712598.2013.758711. Epub 2013 Jan 4. PMID 23286823
- [Background] Di Pierro F, Colombo M, Zanvit A, Rottoli AS. Positive clinical outcomes derived from using Streptococcus salivarius K12 to prevent streptococcal pharyngotonsillitis in children: a pilot investigation. Drug Healthc Patient Saf. 2016 Nov 21;8:77-81. doi: 10.2147/DHPS.S117214. eCollection 2016. PMID 27920580
- [Background] Di Pierro F, Colombo M, Giuliani MG, Danza ML, Basile I, Bollani T, Conti AM, Zanvit A, Rottoli AS. Effect of administration of Streptococcus salivarius K12 on the occurrence of streptococcal pharyngo-tonsillitis, scarlet fever and acute otitis media in 3 years old children. Eur Rev Med Pharmacol Sci. 2016 Nov;20(21):4601-4606. PMID 27874935
- [Background] Di Pierro F, Zanvit A, Nobili P, Risso P, Fornaini C. Cariogram outcome after 90 days of oral treatment with Streptococcus salivarius M18 in children at high risk for dental caries: results of a randomized, controlled study. Clin Cosmet Investig Dent. 2015 Oct 3;7:107-13. doi: 10.2147/CCIDE.S93066. eCollection 2015. PMID 26491371